CLINICAL TRIAL: NCT00523315
Title: A Prospective Observational Study of Compliance in the Patients Receiving Aromatase Inhibitor as an Adjuvant Therapy in Postmenopausal Early Breast Cancer
Brief Title: APOLLO(Aromatase Inhibitor Patient cOmpLiance Program With qoL Questionaire)
Acronym: APOLLO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Other Study IDs: NIS-OKR-ARI-2007/1
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: Aromatase Inhibitor; Breast Cancer; compliance; Naturalistic; Observational
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe patients' compliance of taking Aromatase Inhibitor as an adjuvant treatment in the postmenopausal, early breast cancer as seen under current practice

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients with early breast cancer who are scheduled to receive first-line adjuvant endocrine therapy with aromatase inhibitor under the routine clinical practice
* Histologically or cytologically proven to be HR+(ER or PR +)
* Postmenopausal woman, defined as a woman fulfilling any of the following criteria(by the local guideline):

  * Age >= 50 years
  * Age < 50 years with amenorrhoea > 12 months and an intact uterus
  * FSH levels within postmenopausal range (over 30-40 IU/ml), or
  * Having undergone a bilateral oophorectomy.
  * No other concomitant endocrine therapy such as estrogen therapy or selective estrogen receptor modulators

Exclusion Criteria:

* Recurrence of breast cancer
* Known hypersensitivity to aromatase inhibitor or to any of the excipients
* Any severe concomitant condition which makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the trial protocol
* Previous inclusion in the present study
* Participation in a clinical study during the last 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Surgery or Department of Hemato-oncology in 36 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 862 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, Study Director — AstraZeneca Korea
Locations (19):
- South Korea (19):
  - Research Site, Cheonan-si, Chuncheongnam-do
  - Research Site, Kangnung-si, Gangwon-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Jinju, Gyeongsangnam-do
  - Research Site, Anyang-si, Gyunggi-do
  - Reserach Site, Euijungbu-si, Gyunggi-do
  - Research Site, Seongnam, Gyunggi-do
  - Research Site, Suwon, Gyunggi-do
  - Research Site, Iksan-si, Jeollabuk-do
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Daejoen
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Ulsan